CLINICAL TRIAL: NCT07268105
Title: Flange Fitting for NICU Pumping Parents to Explore Improved Milk Production and Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HP-00114021; HP-00114021 (Other: University of Maryland, Baltimore)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Human Milk/Breastfeeding; Breast Pumping
Keywords: breast pump; human milk
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: The intervention is the type of fitting provided for using the pump. Usual fitting versus the FLANGEFITs protocol.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/usual care (Active Comparator): Pumping people will be provided the usual education and flange fitting procedures.
  Interventions: Other: The intervention is an educational intervention using the FLANGEFits protocol in the NICU. This protocol has only been used previously in the community.
- Intervention group (Experimental): This groups will receive the FLANGEFITS protocol.
  Interventions: Other: The intervention is an educational intervention using the FLANGEFits protocol in the NICU. This protocol has only been used previously in the community.

INTERVENTIONS:
Other: The intervention is an educational intervention using the FLANGEFits protocol in the NICU. This protocol has only been used previously in the community. — The intervention is an educational intervention using the FLANGEFits protocol in the NICU. This protocol has only been used previously in the community.

SUMMARY:
Increasing evidence for an effective method of flange fitting will allow lactation consultants to better advocate for the supplies and training needed to properly fit flanges for this population, hopefully leading to increased milk output and improved experience for parents. Flanges are the part of the pump that fits over the breast and through suction, pulls on the nipple to extract the milk. Recent research showed that a new method of breast pump flange fitting, the Flange FITS TM Guide sizing method, increased milk output and improved the breast milk pumping experience for parents of healthy, term babies.

We hypothesize that the Flange FITS TM Guide sizing method will be effective in NICU parents, a population that has not been explored in current research.

We are conducting a randomized control trial to explore whether the Flange FITS process is better than the standard (manufacturers instructions) for breastpump flange fitting for new parents who are pumping their milk for their newborns in the NICU. We will randomize (1:1) participants to either the new type of flange fitting (Flange FITS) or usual standard care. The study team will assist the pumping parent participant with flange fitting according to their group. This study will ask the pumping parent participants for information about their child and their experience with pumping, and requests that they record the weight of their breast milk after each pump while in the study. The participants already have the pumps and flanges as part of their standard of care. The researchers will provide participants with a scale to weight their breastmilk after each pump while int he study. The researchers will not go into the medical record to retrieve information for the purposes of the study; all information collected for the study will come from the pumping parent participant.

DETAILED DESCRIPTION:
Recent research shows that a new method of breast pump flange fitting, the Flange FITS TM Guide sizing method, increased milk output and improved the breast milk pumping experience for parents of healthy, term babies. https://www.babiesincommon.com/flange-fits-guide Increasing evidence for an effective method of flange fitting will allow lactation consultants to better advocate for the supplies and training needed to properly fit flanges for this population, hopefully leading to increased milk output and improved experience for parents.

In this study we will 1:1 randomize lactating people with neonates in the NICU to the experimental group (Flange FITS Guide sizing method) or the control group (flange manufacturers sizing guide).

The investigators hypothesize that the Flange FITS TM Guide sizing method will be effective in NICU parents, a population that has not been explored in current research.

Aims:

1. Determine if there is an increase in breastmilk production with pumping using the Flange FITS TM Guide sizing method.
2. Determine in there is an increase in comfort with breastfeeding, breastfeeding satisfaction, length of pumping with the use of the Flange FITS TM Guide sizing method.

ELIGIBILITY:
Inclusion Criteria:

* Have newborn in NICU
* Using a breast pump Ability to pump 6-8 times a day

Exclusion Criteria:

* Not using a breast pump No newborn in the NICU

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Weight of milk | Maximum participation is 3 weeks
  The weight of the milk will be collected. A food grade scale will be used.

SECONDARY OUTCOMES:
Pumping satisfaction | Maximum participation in 3 weeks.
  Satisfaction with use of the pump will be collected with a validated measure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a small internal grant. We also need to protect the privacy of participants. We plan to publish results.

REFERENCES:
- [Result] Purdy IB, Singh N, Le C, Bell C, Whiteside C, Collins M. Biophysiologic and social stress relationships with breast milk feeding pre- and post-discharge from the neonatal intensive care unit. J Obstet Gynecol Neonatal Nurs. 2012 May-Jun;41(3):347-57. doi: 10.1111/j.1552-6909.2012.01368.x. PMID 22834882
- [Result] Alves E, Rodrigues C, Fraga S, Barros H, Silva S. Parents' views on factors that help or hinder breast milk supply in neonatal care units: systematic review. Arch Dis Child Fetal Neonatal Ed. 2013 Nov;98(6):F511-7. doi: 10.1136/archdischild-2013-304029. Epub 2013 Jul 18. PMID 23867708
- [Result] Anders LA, Robinson K, Ohlendorf JM, Hanson L. Unseen, unheard: a qualitative analysis of women's experiences of exclusively expressing breast milk. BMC Pregnancy Childbirth. 2022 Jan 21;22(1):58. doi: 10.1186/s12884-022-04388-6. PMID 35062895
- [Result] Meek JY, Noble L; Section on Breastfeeding. Policy Statement: Breastfeeding and the Use of Human Milk. Pediatrics. 2022 Jul 1;150(1):e2022057988. doi: 10.1542/peds.2022-057988. PMID 35921640
- [Result] Lau CYK, Lok KYW, Tarrant M. Breastfeeding Duration and the Theory of Planned Behavior and Breastfeeding Self-Efficacy Framework: A Systematic Review of Observational Studies. Matern Child Health J. 2018 Mar;22(3):327-342. doi: 10.1007/s10995-018-2453-x. PMID 29427014